CLINICAL TRIAL: NCT03518567
Title: Behavioral Economic Analysis of Demand for Marijuana
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brown University (Other)
Responsible Party: Principal Investigator, Elizabeth Aston, Assistant Professor, Brown University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: #1502001185
Record Dates: First submitted 2018-04-09; First posted 2018-05-08 (Actual); Results first posted 2024-02-12 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Marijuana Smoking
MeSH Terms: conditions — Marijuana Smoking | interventions — Dronabinol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- High THC dose (6% THC) (Experimental): Smoked marijuana cigarettes (High THC dose [6% THC])
  Interventions: Drug: Smoked marijuana cigarettes: High THC dose (6% THC)

INTERVENTIONS:
Drug: Smoked marijuana cigarettes: High THC dose (6% THC) — Smoked marijuana cigarettes (High THC dose [6% THC])

SUMMARY:
This laboratory study will employ a multi-session experimental design to examine the behavioral economic demand for marijuana, by studying effect of marijuana administration (High THC) on demand for marijuana, and marijuana smoking topography. The study will recruit 100 non-treatment seeking marijuana users who smoke marijuana at least twice weekly.

DETAILED DESCRIPTION:
This laboratory study will employ a multi-session experimental design to examine craving for marijuana, the effect of marijuana administration (High THC) on behavioral economic demand for marijuana, and marijuana smoking topography. The study will recruit 100 non-treatment seeking marijuana users who smoke marijuana at least twice weekly. The relationship between hypothetical and actual demand for marijuana will be examined. We will also investigate relationship between demand for marijuana and indices of marijuana smoking topography. The study will recruit 100 non-treatment seeking marijuana users who smoke marijuana at least twice weekly to obtain a final sample of 85 with complete data (15% of attrition). Participants will be tested at a baseline session and during two experimental sessions (an ad libitum marijuana smoking session and a marijuana smoking topography session). This study will confirm the utility of the hypothetical marijuana purchase task as a reliable and valid tool for assessing behavioral economic marijuana demand.

ELIGIBILITY:
Inclusion Criteria:

* marijuana use at least 8 times in the past month on average and at least monthly for the past 6 months
* English-speaking
* negative urine toxicology screen for drugs other than marijuana
* non-treatment seeking
* purchase of marijuana at least twice in the past 6 months to confirm familiarity with the construct to be measured

Exclusion Criteria:

* positive pregnancy test
* nursing
* inability to use contraception during the study
* poor physical health
* positive breath alcohol concentration
* diagnosis of a current affective disorder, psychosis, and panic disorder
* self-report of past serious adverse reaction to marijuana
* current psychotropic drug use
* smoking more than 20 tobacco cigarettes per day
* inability to abstain from marijuana for 15 hours
* body mass index outside 18.5-30 kg/m2 range

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 133 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2021-05-24 (Actual); Study Completion 2021-05-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Aston, PhD, Principal Investigator — Brown University
Locations (1):
- Brown University, Providence, Rhode Island, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | High THC Dose (6% THC)
Started | 133
Completed Baseline | 114
Completed Session 1 | 101
Completed Session 2 | 72
Completed (This is the number of participants who completed Baseline, Session 1, and Session 2.) | 72
Not Completed | 61

BASELINE CHARACTERISTICS:
Arm/Group | High THC Dose (6% THC)
Number analyzed (Participants) | 114
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.6 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50
  Male | 64
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20
  Not Hispanic or Latino | 94
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 10
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 19
  White | 72
  More than one race | 9
  Unknown or Not Reported | 4

OUTCOME MEASURES:

1. Primary Outcome: Validity of the Marijuana Purchase Task (MPT)
Description: The Marijuana Purchase Task will be used to collect data on marijuana demand. Participants indicate how much marijuana they would purchase at varying levels of price (e.g., free - $60). Indices of marijuana demand are derived from the task and used to determine the relative value of marijuana for each participant. Hits purchased on the MPT will correspond with actual number of hits purchased and smoked in the laboratory. Primary outcome is percentage of participants who purchased and smoked exactly what they said they would.
Time Frame: Duration of the experimental session (i.e., 60 minutes)
Population: All participants who completed Session 1 (n=101), reported purchasing at least 1 hit from a cannabis joint at their randomly selected price-point on the Marijuana Purchase Task (n=90), and chose to smoke during the Session (n=86) were included in the analysis. Outcome corresponds to percentage of participants who smoked exactly what they said they would.
Measure: Number; unit: percentage of participants
Arm/Group | High THC Dose (6% THC)
Number analyzed (Participants) | 86
percentage of participants | 63
Statistical Analysis 1: Comparison: High THC Dose (6% THC); Test type: Superiority; p = .00000004, Regression, Linear; hits purchased on the MPT predicting hits actually purchased and smoked in the laboratory. covariate: baseline total individual income; Slope = 0.78

2. Secondary Outcome: Change in Marijuana Craving Questionnaire (MCQ)
Description: Subjective marijuana craving was assessed via a 10-item Marijuana Craving Questionnaire. Participants were asked to respond to items according to how they were thinking or feeling "right now," and MCQ items were rated on a 1 = "strongly disagree" to 7 = "strongly agree" scale, with higher scores indicating greater subjective marijuana craving, and summed to yield a total craving score. Total craving score was used in analyses.
Time Frame: The MCQ will be administered pre- and post- marijuana smoking during the experimental session, up to 6 hours
Population: All participants who completed Session 1 (n=101), reported purchasing at least 1 hit from a cannabis joint at their randomly selected price-point on the Marijuana Purchase Task (n=90), and chose to smoke during the Session (n=86) were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on the MCQ
Arm/Group | High THC Dose (6% THC)
Number analyzed (Participants) | 86
units on the MCQ | -0.75 (1.09)
Statistical Analysis 1: Comparison: High THC Dose (6% THC); Test type: Superiority; p = .000000009, t-test, 2 sided; Mean Difference (Final Values) = -0.75, Standard Deviation 1.09

3. Secondary Outcome: Marijuana Smoking Topography
Description: Indices of Marijuana Smoking Topography will be obtained during the experimental session. Participants will smoke marijuana through a smoking topography device. The outcome measure is number of puffs.
Time Frame: Marijuana smoking topography indices will be collected during the 1-hour ad libitum marijuana smoking topography experimental session.
Population: Participants who completed Session 2 with usable smoking topography data.
Measure: Mean (Standard Deviation); unit: puffs
Arm/Group | High THC Dose (6% THC)
Number analyzed (Participants) | 67
puffs | 29 (13.7)
Statistical Analysis 1: Comparison: High THC Dose (6% THC); Test type: Superiority; p = .87, correlation; Correlation between puffs on the topography device and grams of cannabis used per week; correlation = .02

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | High THC Dose (6% THC)
All-Cause Mortality (participants affected / at risk) | 0/114
Serious Adverse Events (participants affected / at risk) | 0/114
Other Adverse Events (participants affected / at risk) | 0/114

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-10-08): https://cdn.clinicaltrials.gov/large-docs/67/NCT03518567/Prot_SAP_001.pdf
  • Informed Consent Form (2020-10-08): https://cdn.clinicaltrials.gov/large-docs/67/NCT03518567/ICF_000.pdf